CLINICAL TRIAL: NCT00247845
Title: Evaluation of Atazanavir Substitution Intervention (EASI) Study: An Observational Phase IV Study to Evaluate the Impact of Atazanavir Substitution on the Quality of Life and Maintenance of Virologic Suppression in HIV-Infected Patients Intolerant to Current Successful HAART
Brief Title: Evaluation of Atazanavir Substitution Intervention (EASI) Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: P04-0098
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections
Keywords: HIV; Atazanavir; quality of life; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
With the advent of highly active antiretroviral therapy (HAART), it was hypothesized that its consistent use could lead to a cure for HIV infection in as little as three years [Perelson, 1997]. Subsequent research has shown this model to be incorrect [Finzi, 1999]. In addition, long term use of HAART has now been associated with significant metabolic abnormalities, which could lead to unintended morbidity, possibly worse than what one could expect from the progression of untreated HIV-associated immune disease over the same period of time [Carr, 2000]. Accordingly, current recommendations for antiretroviral therapy have become more conservative. It is now suggested that a person with a CD4 count > 350 cells/mm³ may safely delay initiation of HAART [Yeni, 2002].However, for those who still require HAART, the risks of short-term and long-term toxicities remain, even if full virologic suppression is achieved. In this setting, a number of switching strategies have been evaluated (Negredo et al, 2002 & Martinez et al, 2003), mostly involving single drug substitutions of a protease inhibitor (PI) for a non-nucleoside agent (NNRTI) or abacavir (ABC). In general terms, these hae shown that virologic suppression is usually maintained, with improvement in drug-related side effects, including metabolic toxicities. A number of patients who are currently taking effective HAART are experiencing side effects to one or more of the agents in their regimen that is not severe enough to mandate an immediate change in their regimen, but that is having a measurable effect on their qualify of life. Over time, these effects may have an impact on adherence to therapy and its long-term efficacy. Given the recent availability of ATV (+/-RTV), its once daily administration, low pill count and favourable side effect profile, it is being used in clinical practice as part of single drug substitution strategies in patients exhibiting a maximal response to HAART. There is a clear need to examine this practice in a systematic manner to document its occurrence, efficacy and safety.

We hypothesize that, in patients with maximal virologic suppression on a double class regimen (including two NRTIs and an NNRTI or a PI, boosted with RTV or not), and in whom a decision has been made to implement a single drug substitution of the NNRTI or PI for ATV (+/-), this will lead to an improvement in objectively measured quality of life without any negative impact on the virologic efficacy of the regimen.

DETAILED DESCRIPTION:
This will be a single arm observational study to include 100 subjects. After a clinical decision is made to implement a single drug substitution to ATV +/- RTV, there will be an initial screening visit, at which time the study will be presented to the patient and informed consent for participation will be obtained. A number of evaluations (including blood tests) will be completed to definitively assess a subject's eligibility to participate in this protocol. The patients will continue on their current therapy and will return within the next 14 days for an enrollment visit to review the blood test results and definitively confirm study eligibility. In particular, we will ascertain the continued presence of the side effect/toxicity motivating consideration of a change in therapy. This being down, the quality of life questionnaires (MOS-HIV and ASDM) will be administered for the first time. Once again, the patient will continue on their current HAART and return within the next 14 days for a baseline visit at which time the quality of life questionnaires (MOS-HIV and ASDM) will be administered once again, the results being averaged with those obtained at the time of the enrollment visit, this serving as a more rigorous evaluation of the patient's current status. The patient could be withdrawn from the study if the side effect/toxicity motivating consideration of a change in therapy is no longer present. At this baseline visit, all patients will switch the PI or NNRTI component of their regimen to ATV (+/- RTV). The decision to use boosted or unboosted ATV in this protocol will be left to the discretion of the treating physician. All patients will be receiving ATV (+/- RTV) with food. The dose of the unboosted ATV will be 300 mg (2 capsules, 150mg each) plus RTV (1 capsule, 100 mg). The patients will then be seen in follow up at weeks 4, 12, 24, 32, and 48 after the baseline visit. They will continue on their new therapy (including ATV +/- RTV) for this entire period of observation. Changes in the NRTI backbone will be permitted without constituting a study endpoint, while changes in the ATV +/- RTV that may be required for reasons of efficacy or toxicity will constitute such an endpoint, leading to a patient's withdrawal from the study. At each study visit, the quality of life questionnaires (MOS-HIV and ASDM) will be administered. The results will be compared to the mean results obtained at the enrollment and baseline visits, with each individual participant serving as his/her own control. Measures of adherence to HAART, CD4 cell counts and HIV plasma viral load will also be obtained at each study visit, and will constitute secondary study endpoints.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older; a confirmed diagnosis of HIV infection; 2 consecutive HIV RNA levels <50 copies/mL with the most recent being within the past 3 months; have been on the same HAART regimen for the past 3 months; have side effects to their current antiretroviral medications that warrant a consideration of a change in therapy. There must be a clinical suspicion by the investigator that these side effects are attributable to either the PI or the NNRTI component of the regimen; Have agreement between the treating physician and the patient that a single drug substitution to ATV +/- RTV will be proposed, independent of participation in the study; be able to provide written informed consent and complete the quality of life instruments and, in the opinion of the investigator, comply in every other way with the requirements of the study protocol.

Exclusion Criteria:

Exclusion criteria: Have received investigational drug within 30 days prior to the baseline visit of the study; if female, be pregnant or breast-feeding; have an acute illness, including an acute opportunistic infection; have grade 3-4 laboratory abnormalities on any of the following parameters: CBC, ALT, AST, GGT, LDH, bilirubin, amylase, and alkaline phosphatase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age or older with a confirmed diagnosis of HIV infection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-07; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Conway, MD, Principal Investigator — University of British Columbia
Locations (5):
- Canada (5):
  - Downtown Infectious Diseases Clinic,, Vancouver, British Columbia
  - Oak Tree Clinic, Vancouver, British Columbia
  - Pender Community Health Center, Vancouver, British Columbia
  - Vancouver General Hospital Clinic, Vancouver, British Columbia
  - Cool-Aid Society in Victoria, Victoria, British Columbia